CLINICAL TRIAL: NCT03708042
Title: A Phase Ⅲ Trial to Compare Efficacy and Safety of Definitive Chemoradiation VS Neoadjuvant Chemoradiation Plus Surgery in Patients Who Achieved Clinical Complete Response After Neoadjuvant Treatment for Locally Advanced Esophageal Cancer
Brief Title: A Study to Compare Efficacy and Safety of DRT VS CRT Plus Surgery in Patients Who Achieved CCR for Esophageal Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other); Sun Yat-sen University (Other); Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESO20181012
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Stage II Esophageal Cancer; Stage III Esophageal Cancer
Keywords: Neoadjuvant Chemoradiation; Definitive Chemoradiation; Clinical complete response
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Definitive Radiochemotherapy (Experimental): Radiotherapy,IMRT, 60Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day.
  Interventions: Combination Product: Definitive Radiochemotherapy
- Neoadjuvant Radiochemotherapy (Active Comparator): Radiotherapy,IMRT, 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day; Receive radical surgery 4 to 6 weeks later.
  Interventions: Combination Product: Neoadjuvant Radiochemotherapy

INTERVENTIONS:
Combination Product: Definitive Radiochemotherapy — Radiotherapy,IMRT, 60Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day
  Arms: Definitive Radiochemotherapy
Combination Product: Neoadjuvant Radiochemotherapy — Concurrent Radiochemotherapy: Radiotherapy,IMRT, 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2) 1st/8th/15th/22nd day; Receive radical surgery 4 to 6 weeks later.
  Arms: Neoadjuvant Radiochemotherapy

SUMMARY:
Neoadjuvant chemoradiotherapy(Neo-CRT) plus surgery has been regarded as a standard of care for patients with resectable locally advanced esophageal cancer. Many studies suggest that definitive Radiochemotherapy(CRT) has similar efficacy as neoadjuvant chemoradiotherapy plus surgery for esophageal cancers who respond to chemoradiation. Herein, a single center prospective randomized phase Ⅲ multicenter clinical trial will be carried out to compare efficacy and safety of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection in patients who achieved clinical complete response (CCR) after neoadjuvant radiochemotherapy for resectable locally advanced esophageal cancer.

DETAILED DESCRIPTION:
1. Compare progression-free survival (PFS) and overall survival (OS) of definitive radiochemotherapy versus(VS) neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant treatment;
2. Compare the toxic and side effects of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete remission after neoadjuvant treatment;
3. Compare the relationship and consistency between pathological complete response of endoscopic biopsy specimens after neoadjuvant treatment and pathological complete response of surgical specimens in neoadjuvant radiochemotherapy plus radical resection group;
4. Assess impact of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection on quality of life of patients.
5. Clinical Complete Response After Neoadjuvant Treatment: Endoscope biopsy pathologic diagnosis indicate pathologic complete response after Neoadjuvant treatment; upper gastrointestinal/chest CT and symptom assessment indicate major response after Neoadjuvant treatment (Concurrent Radiochemotherapy: Radiotherapy, Intensity Modulation Radiation Therapy(IMRT), 40Gy; Chemotherapy, Docetaxel （25mg/m2）+Cisplatin (25mg/m2), 1st/8th/15th/22nd day

ELIGIBILITY:
Inclusion Criteria:

1. Thoracic esophageal cancer patients or esophagocardial cancer patients, with locally advanced resectable tumor, clinically identified before treatment as T1-3N+M0 according to UICC(International Union Against Cancer) TNM(primary tumor, regional nodes, metastasis) Classification of Malignant Tumours, 8th ed.
2. Untreated patients who have not received any antitumor therapy
3. Life expectancy >6 months
4. Age: 18-70 years
5. White blood cell count ≥4.0×109/l, ANC(absolute neutrophil count) ≥1.5×109/l, thrombocyte count ≥1011/l, hemoglobin ≥90 g/l; normal liver and kidney functions
6. WHO PS(Performance Status): 0-1
7. Patients who understood the study and gave signed informed consent

Exclusion Criteria:

1. Patients who have already received antitumor therapy, including chemotherapy, radiotherapy or surgery;
2. Patients who suffered from hemorrhage or complicated hemorrhage;
3. Other uncontrollable patients who are not suitable for surgery;
4. Female patients in pregnancy or lactation;
5. Patients who agree without acknowledgement due to psychic, family or social factors;
6. Patients who suffered from peripheral neuropathy, with CTC grade ≥2;
7. Patients who ever suffered from other types of malignant tumor other than esophagus cancer;
8. Patients who have diabetes history over 10 yrs and blood glucose level is not satisfyingly controlled;
9. Patients who suffer from serious malfunction of heart, lung, liver or kidney, hemotopathy, immune system disease or cachexia and therefore can't tolerate chemotherapy or surgery;
10. Others.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 years
  Compare overall survival of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant radiochemotherapy

SECONDARY OUTCOMES:
Progression-free survival | 3 years
  Compare progression-free survival of definitive radiochemotherapy versus neoadjuvant radiochemotherapy plus radical resection for esophageal cancer patients who achieved clinical complete response after neoadjuvant radiochemotherapy
Number of Participants With Abnormal Laboratory Values and/or Adverse Events That Are Related to Treatment | 5 years
  grade 3 or 4 toxicity of leukocytes, febrile neutropenia, thrombocytes, hemoglobin, nausea/vomiting, diarrhea, stomatitis, esophagitis, cardiovascular.
Comparison of pathological diagnosis between specimens of endoscopic biopsy and surgically resected in esophageal cancer | 3 years
  In the group of neoadjuvant radiochemotherapy plus surgery, we will compare the pathological diagnosis between specimens of endoscopic biopsy after neoadjuvant treatment and surgically resected.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Wang, PHD & MD, Study Chair — Department of Radiation Oncology, Tianjin Medical University Cancer Hospital

IPD SHARING:
Plan to Share IPD: No